CLINICAL TRIAL: NCT01598532
Title: Treatment of Cognitive Dysfunction in Mild TBI With Transcranial Light Emitting Diodes- An Open Protocol, Pilot Study
Brief Title: Effects of LEDs on Memory in TBI Patients
Acronym: LED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Ross D. Zafonte, MD, Vice President Medical Affairs, Research and Education Spaulding Rehabilitation Network, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-P-001552
Record Dates: First submitted 2012-05-04; First posted 2012-05-15 (Estimated); Results first posted 2016-08-22 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Traumatic Brain Injury
Keywords: mild traumatic brain injury; mild TBI; mTBI
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transcranial LED Treatment (Experimental): All study subjects received treatment during 6-Week period (3x per week) for a total of 18 Transcranial LED Treatments using the MedX Health Phototherapy (light). Each session was 30 minutes in duration.
  Interventions: Device: MedX Health Phototherapy (light therapy)

INTERVENTIONS:
Device: MedX Health Phototherapy (light therapy) — The treatment period is 6 weeks (3x per week) for a total of 18 Transcranial LED treatments. Each treatment session is 30 minutes each.

SUMMARY:
The purpose of the study is to investigate whether transcranial, high-intensity LED placed on the scalp can improve working memory in people who have sustained a concussion with lingering effects or a mild brain injury.

DETAILED DESCRIPTION:
This is a four month, outpatient, single center study investigating whether transcranial, high intensity LED applied outside the skull can improve frontal lobe executive function and working memory in participants with chronic, mild Traumatic Brain Injury (TBI), with or without mild posttraumatic stress disorder (PTSD), due to closed head injury.

Participants will sign the Informed Consent Form(ICF) before Neuropsychological Screening test are administered. If the participant's neuropsychological screening test scores meet the Inclusion/Exclusion criteria and the participant meets the other Inclusion/Exclusion criteria, then he/she will be tested again on the tests that are part of the Neuropsychological Outcome Measures, the week before the Transcranial LED treatments, and during the week after the last LED treatment and again at one and two months after the last LED treatment. Treatment with Transcranial LED will be for 6 weeks. Participants will be treated three times per week: Monday, Wednesday and Friday. A total of 18 Transcranial LED treatments will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, Ages 18-65
* sustained a mild traumatic brain injury(mTBI) at least 6 months ago
* mTBI is defined as < 30 minutes loss of consciousness and <30 minutes, post trauma amnesia
* since the injury patient continues having problems with memory and thinking ability

Exclusion Criteria:

* Younger than 18 or older than 65
* mTBI occured less than 6 months ago
* moderate to severe Traumatic Brain Injury (TBI)
* non-closed head injury
* presence of craniotomy, craniectomy, or ventriculoperitoneal shunt
* Non-English speaking subjects - Neuropsychological Tests only in English
* Neuropsychological Screening Test Scores not at least 2 SD below norm on one of the neuropsychological tests or not 1 SD below norm on at least two of the tests administered during screening)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross D Zafonte, DO, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hashmi JT, Huang YY, Osmani BZ, Sharma SK, Naeser MA, Hamblin MR. Role of low-level laser therapy in neurorehabilitation. PM R. 2010 Dec;2(12 Suppl 2):S292-305. doi: 10.1016/j.pmrj.2010.10.013. PMID 21172691
- [Result] Naeser MA, Saltmarche A, Krengel MH, Hamblin MR, Knight JA. Improved cognitive function after transcranial, light-emitting diode treatments in chronic, traumatic brain injury: two case reports. Photomed Laser Surg. 2011 May;29(5):351-8. doi: 10.1089/pho.2010.2814. Epub 2010 Dec 23. PMID 21182447
- See also: Department of Physical Medicine and Rehabilitation at Spaulding Hospital - Research — http://pmr.hms.harvard.edu/pages/10/119/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the study began in April 2010. Potential subjects were recruited through several different methods - Spaulding Rehabilitation Hospital outpatient clinic, advertisements in local area newspapers, Brain Injury Association of MA and other area organizations that provide services to TBI survivors, flyers, on-line and social media.
Pre-assignment Details: 22 study subjects signed the consent but only 11 completed the study. The 11 that did not completed the study either did not meet the inclusion criteria at Screening or were lost to follow-up after they screened for the study.
Groups:
- Transcranial LED Treatment: Population was Males and Females, ages 18 to 65 years who sustained a mild traumatic brain injury at least 6 months prior to study participation. All study subjects received treatment during 6-Week period (3x per week) for a total of 18 Transcranial LED Treatments using the MedX Health Phototherapy (light). Each session was 30 minutes in duration.
Period: Overall Study
Arm/Group | Transcranial LED Treatment
Started | 22
Completed | 11
Not Completed | 11
Not completed — Lost to Follow-up | 3
Not completed — Did not meet inclusion criteria | 8

BASELINE CHARACTERISTICS:
Population: Population was Males and Females, ages 18 to 65 years who sustained a mild traumatic brain injury at least 6 months prior to study participation
Groups:
- Transcranial LED Treatment: All study subjects received LED treatment during 6-Week period (3x per week) for a total of 18 Transcranial LED Treatments using the MedX Health Phototherapy. Each session was 30 minutes in duration. Neuropsychological testing was administered at the following time points: within 1 week of the first LED treatment and within 1 week, 1 month & 2 months following the last LED treatment.
  The neuropsychological testing included: 1)Stroop test, 2) California Verbal Learning Test-II (CVLT- II), Short Delay Free & Cued Recall, Long Delay Free & Cued Recall, 3) Delis-Kaplan Executive Function (D-KEF) -Trails Test, 4) Controlled Oral Word Association Test (FAS), & 5) Digit Span, Forwards & Backwards.
  The following tests were not analyzed due to collinearity with other measures (r > .8): Short Delay Free & Cued Recall, Long Delay Cued Recall, & Delis-Kaplan Executive Function (D-KEF) -Trails Test.
Arm/Group | Transcranial LED Treatment
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Time Post TBI [Mean (Standard Deviation); unit: years post TBI] — This calculates the time elapsed since injury
  years post TBI | 3.12 (2.50)
Years of Education [Mean (Standard Deviation); unit: Years of Education] — Numbers of years of education
  Years of Education | 15.72 (2.97)

OUTCOME MEASURES:

1. Primary Outcome: Stroop Test for Executive Function - Trial 3 - Inhibition
Description: Stroop Test for Executive Function - Trial 3 (D-KEFS) - Inhibition measures executive function, inhibition that has been converted to Z-score, # of Standard Deviation units. Higher Mean scores equals better outcomes.
Time Frame: Baseline and 1-Week, 1-month and 2-months after final LED Treatment
Population: All participants enrolled in the Transcranial LED Treatment Group
Measure: Mean (Standard Deviation); unit: # of SD units
Arm/Group | Transcranial LED Treatment
Number analyzed (Participants) | 11
# of SD units
  Pre-test data | -0.7407 (1.1561)
  1 Week post test data | .036 (.7407)
  1 Month post test data | .718 (1.0133)
  2 Months post test data | .815 (.9499)
Statistical Analysis 1: Comparison: Transcranial LED Treatment; linear trend over time for the effect of LED treatments; Test type: Superiority or Other; p < 0.004, ANOVA; Univariate, one-way, repeated measure ANOVA with trend analysis

2. Primary Outcome: Stroop Test for Executive Function - Trial 4 Inhibition Switching
Description: Stroop Test for Executive Function - Trial 4 (D-KEFS) Inhibition Switching that has been converted to Z-score, # of Standard Deviation units. Higher Mean scores equals better outcomes.
Time Frame: Baseline and 1-Week, 1-Month and 2-Months after the Final LED Treatment
Population: All participants enrolled in Transcranial LED Treatment Group
Measure: Mean (Standard Deviation); unit: # of SD Units
Arm/Group | Transcranial LED Treatment
Number analyzed (Participants) | 11
# of SD Units
  Pre-test data | -1.050 (1.1058)
  1 week post test data | -0.100 (1.3994)
  1 Month post test data | .553 (1.167)
  2 Month post test data | .854 (1.3544)
Statistical Analysis 1: Comparison: Transcranial LED Treatment; linear trend over time for the effect of LED treatments; Test type: Superiority or Other; p < 0.003, ANOVA; Univariate, one-way, repeated measure ANOVA with trend analysis

3. Primary Outcome: California Verbal Learning Test-II (CVLT-II) Total, Trials 1-5
Description: California Verbal Learning Test-II (CVLT-II) Total, Trials 1 - 5 measures word recall on trials 1-5 that has been converted to Z-score, # of Standard Deviation units. Higher Mean scores equals better outcomes.
Time Frame: Baseline and 1-Week, 1-Month and 2-Months after Final LED Treatment
Population: All participants enrolled in Real Intervention Group
Measure: Mean (Standard Deviation); unit: # of SD Units
Groups:
- Transcranial LED Treatment: Population was Males and Females, ages 18 to 65 years who sustained a mild traumatic brain injury at least 6 months prior to study participation. All study subjects received treatment during 6-Week period (3x per week) for a total of 18 Transcranial LED Treatments using the MedX Health Phototherapy (light and laser). Each session was 30 minutes in duration.
Arm/Group | Transcranial LED Treatment
Number analyzed (Participants) | 11
# of SD Units
  Pre-test Data | -.409 (.7687)
  1 Week post test data | .364 (.809)
  1 Month post test data | .630 (.7015)
  2 Month post test data | .780 (.9724)
Statistical Analysis 1: Comparison: Transcranial LED Treatment; linear trend over time for effect of LED treatments; Test type: Superiority or Other; p < 0.003, ANOVA; Univariate, one-way, repeated measure ANOVA with trend analysis

4. Primary Outcome: California Verbal Learning Test-II (CVLT-II) Long Delay Free Recall
Description: California Verbal Learning Test-II (CVLT-II) Long Delay Free Recall measures word recall after a 20 minute delay that has been converted to Z-score, # of Standard Deviation units. Higher Mean scores equals better outcomes.
Time Frame: Baseline and 1-Week, 1-Month and 2-Months after final LED Treatment
Population: All participants enrolled in Transcranial LED Treatment Group
Measure: Mean (Standard Deviation); unit: # of SD Units
Arm/Group | Transcranial LED Treatment
Number analyzed (Participants) | 11
# of SD Units
  Pre-test data | -1.136 (1.4334)
  1 Week post test data | -0.136 (1.1851)
  1 Month post test data | -0.200 (1.249)
  2 Month post test data | 0.050 (1.15)
Statistical Analysis 1: Comparison: Transcranial LED Treatment; linear trend over time for the effects of LED treatments; Test type: Superiority or Other; p < 0.006, ANOVA; Univariate, one-way, repeated measure ANOVA with trend analysis

5. Primary Outcome: Controlled Oral Word Association Test (FAS)
Description: Controlled Oral Word Association Test (FAS) measures verbal fluency that has been converted to Z-score, # of Standard Deviation units. Higher Mean scores equals better outcomes.
Time Frame: Baseline and 1-Week, 1-Month and 2-Months after final LED Treatment
Population: All participants enrolled in the Transcranial LED Treatment Group
Measure: Mean (Standard Deviation); unit: # of SD units
Arm/Group | Transcranial LED Treatment
Number analyzed (Participants) | 11
# of SD units
  Pre-test data | -.318 (1.54)
  1 Week post test data | .136 (1.45)
  1 Month post test data | .114 (1.58)
  2 Month post test data | .285 (1.38)

6. Primary Outcome: Digit Span, Forwards and Backwards
Description: Digit Span, Forwards and Backwards measures short-term auditory memory and working memory that has been converted to Z-score, # of Standard Deviation units. Higher Mean scores equals better outcomes.
Time Frame: Baseline and 1-Week, 1-Month and 2-Months after final LED Treatment
Population: All participants enrolled in the Transcranial LED Treatment Group
Measure: Mean (Standard Deviation); unit: # of SD units
Arm/Group | Transcranial LED Treatment
Number analyzed (Participants) | 11
# of SD units
  Pre-test data | -.182 (1.45)
  1 Week post test data | .318 (1.31)
  1 Month post test data | .444 (1.42)
  2 Month post test data | .650 (1.52)

ADVERSE EVENTS:
Time Frame: Over a period of 2 years 11 participants were studied with no adverse events
Arm/Group | Transcranial LED Treatment
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
Small sample size & Open Protocol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes